CLINICAL TRIAL: NCT01317654
Title: Study Of The Long Term Outcome Of Tuberculous Meningitis In Vietnamese Adults Treated With Adjunctive Dexamethasone
Acronym: ES
Status: Completed | Type: Observational
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Other Study IDs: ES
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Tuberculosis Meningitis
Keywords: Tuberculosis meningitis
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survivors of TBM trial 2001-2005
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Collection of mortality data at 5 years post trial

SUMMARY:
All patients who were alive at the end of the dexamethasone treatment trial conducted by Oxford University CLinical Research Unit from 2001-2005 (n=340) will be eligible to participate in this long-term follow-up study.

All eligible and consenting patients will undergo an assesment consisting of a simple questionnaire, a clinical examination and a blood test. Data collected will focus on survival, neurological disability and tuberculosis relapse. Data will be collected in individual case record forms and entered into a computer database.

ELIGIBILITY:
Inclusion Criteria:Patients were alive at the end of the dexamethasone study (n=340) will be eligible to participate in this long-term follow-up study Informed consent

Exclusion Criteria:

Patients without informed consent

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Survivors of TBM trial 2001-2005
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Survival | 5 years

SECONDARY OUTCOMES:
Neurological disability | 5 years
Tuberculosis relapse rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Estee Torok, MD, Principal Investigator — Oxford University Clinical Research Unit - Viet Nam

REFERENCES:
- [Derived] Torok ME, Nguyen DB, Tran TH, Nguyen TB, Thwaites GE, Hoang TQ, Nguyen HD, Tran TH, Nguyen TC, Hoang HT, Wolbers M, Farrar JJ. Dexamethasone and long-term outcome of tuberculous meningitis in Vietnamese adults and adolescents. PLoS One. 2011;6(12):e27821. doi: 10.1371/journal.pone.0027821. Epub 2011 Dec 8. PMID 22174748